CLINICAL TRIAL: NCT00988312
Title: Vaccination With Idiotype-KLH Loaded Dendritic Cells. A Phase I Study for Patients With Multiple Myeloma
Brief Title: Dendritic Cells(DC)-Based Id Vaccination in Stage-I Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Carl Gustav Carus (Other)
Responsible Party: Susanne Gretzinger, University Hospital Carl Gustav Carus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyelomVak
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Multiple Myeloma; Plasmocytoma
Keywords: dendritic cells (DC); idiotype (Id); immunotherapy
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- s.c. vaccination (Experimental): vaccine given subcutaneously
  Interventions: Biological: autologous idiotype-protein pulsed dendritic cells
- i.v. vaccination (Experimental): vaccines are given intravenously
  Interventions: Biological: autologous idiotype-protein pulsed dendritic cells

INTERVENTIONS:
Biological: autologous idiotype-protein pulsed dendritic cells — Vaccination with autologous idiotype-protein pulsed dendritic cells on 5 occasions every 4 weeks

SUMMARY:
Patients with stage-I multiple myeloma are treated with a vaccine made from their own immune cells (dendritic cells) and their own myeloma protein. Vaccinations are given on 5 occasions every 4 weeks. The aim is to induce an immune reaction against the malignant myeloma cells in order to slow down or cure the disease.

ELIGIBILITY:
Inclusion Criteria:

* multiple myeloma
* stage I (Salmon & Durie)
* no cytoreductive pre-treatment

Exclusion Criteria:

* myeloma stages II-III
* asecretory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-03; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Specific T-cell proliferation/cytokine secretion

SECONDARY OUTCOMES:
number of T cells | pre and post vaccination
monoclonal protein | pre and post vaccination
plasmacells in bone marrow | pre and post vaccination
vital signs | pre and post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Gretzinger, MD, Principal Investigator — University Hospital Dresden
Locations (1):
- University Hospital Dresden, Dresden, Germany